CLINICAL TRIAL: NCT02639832
Title: A Pilot Surveillance Study to Monitor Natural Killer Cells and Circulating Tumor Cells in Women With Previously Treated Non-metastatic Triple Negative Breast Cancer and Women With Previously Treated Non-metastatic Breast Cancer With a Confirmed BRCA Mutation.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cynvenio Biosystems (Industry)
Responsible Party: Sponsor
Other Study IDs: SAIRB-15-0060
Record Dates: First submitted 2015-12-10; First posted 2015-12-24 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Triple Negative Breast Cancer; Natural Killer Cells; BRCA Mutation
Keywords: Triple Negative Breast Cancer; Breast Cancer; Natural Killer Cells; BRCA Mutation
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: LiquidBiopsy®, NK VueTM — The LiquidBiopsy® device will test for cells with tumor cell markers in blood. The genetic sequence of DNA recovered samples will be studied. Using NK VueTM researchers will test for NK cell activity.

SUMMARY:
The purpose of this research study is:

* To test blood for the presence of tumor derived circulating tumor cells (CTCs) or circulating tumor DNA (ctDNA) using an investigational medical device called the LiquidBiopsy®. Using the LiquidBiopsy® platform, recovered cells or DNA can also be investigated to obtain genetic information that may be useful to treating physicians in understanding disease.
* To test blood for natural killer cells (NK cells), which are part of the body's natural immune defense against tumors. A device called the NK VueTM Kit will be used for this test.

The LiquidBiopsy® is a new investigational device. An investigational device is one that is not approved by the United States Food and Drug Administration (FDA). The NK VueTM Kit is an investigational device in the United States but is approved in Canada and South Korea as a class II device.

If a tumor is present, very tiny numbers of tumor cells or the contents of these tumor cells can get dislodged from the tumor and swept into the bloodstream. The LiquidBiopsy® device is able to purify the tiny numbers of tumor cells or ctDNA in the blood. Even if a tumor is too small to be found by other means such as an x-ray, it is possible that ctDNA or CTCs may be found in the blood. Genetic information can then be recovered from these cells or DNA to look for genetic changes that are related to the abnormal growth in a tumor. This will potentially allow researchers to study tumor cells or tumor DNA from a blood sample instead of a biopsy sample. This may influence cancer diagnosis, treatment and drug selection in the future.

NK cells occur naturally in the body and kill tumor cells. This study will measure the activity of the NK cells in blood. A strong correlation between low NK cell activity and increased circulating tumor cells in blood has been reported.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Female.
* Over 18 years of age.
* Previously Treated Non-metastatic Triple Negative Breast Cancer or Women with Previously Treated Non-metastatic Breast Cancer With a confirmed BRCA Mutation who have completed therapy within three years of enrollment in this study.
* Subject may be invited to annual review of the Subject Information and Donation Schedule by email or mail follow up for five years after sampling.
* Subject provides written authorization for use and disclosure of protected health information (PHI).

Exclusion Criteria:

* Any conditions inappropriate for blood drawing.
* Known active viral or bacterial infection at time of blood draw.
* Known HIV, Hepatitis B, or Hepatitis C infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously Treated Non-metastatic Triple Negative Breast Cancer or Breast Cancer with a confirmed BRCA mutation.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Presence of cell free tumor DNA and/or circulating tumor cells from a blood sample in women with Triple Negative Breast Cancer (TNBC) or a confirmed BRCA Mutation who have completed therapy and have no evidence of active disease via LiquidBiopsy. | When NK cell activity is low for up to 3 years.
Natural Killer cell activity levels in women with Triple Negative Breast Cancer and Women with Previously Treated Non-metastatic Breast Cancer or a confirmed BRCA Mutation who have completed therapy and have no evidence of active disease via ELISA assay. | Monthly up to 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Cynvenio Biosystems, Inc., Westlake Village, California, United States